CLINICAL TRIAL: NCT02165917
Title: Randomised, Controlled Clinical Study With Patients With Endometriosis and the Desire to Have Children - Comparison Between Peritoneal Ablation by Excision Only and Excision With the Use of an Adhesionbarrier
Brief Title: Study to Compare Peritoneal Ablation by Excision Only and Excision With the Use of an Adhesion Barrier
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Pius-Hospital Oldenburg (Other)
Responsible Party: Principal Investigator, Prof. Dr. Dr. med. Rudy Leon De Wilde, Professor Dr. Dr. med., Pius-Hospital Oldenburg
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PHDW-003
Record Dates: First submitted 2014-04-15; First posted 2014-06-18 (Estimated); Last update posted 2015-11-03 (Estimated); Status verified 2015-11

CONDITIONS: Endometriosis
Keywords: Endometriosis; Adhesions; Hyalobarrier®; Hyaluronic acid; Antiadhesion agent; Adhesionbarrier; Pregnancy rate
MeSH Terms: conditions — Endometriosis; Tissue Adhesions

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Excision only (Placebo Comparator): Laparoscopic excision of endometriotic lesions followed by 3 month of GnRH-Analogue administration
  Interventions: Procedure: Excision only
- Excision plus hyaluronic acid gel (Active Comparator): Standard Laparoscopic excision of endometriotic lesions plus application of 10 cc of a hyaluronic acid gel (Hyalobarrier® ), followed by 3 month of GnRH-analogue administration
  Interventions: Procedure: Excision plus hyaluronic acid gel

INTERVENTIONS:
Procedure: Excision plus hyaluronic acid gel — Excision of endometriosis foci by laparoscopic standard methods followed by an application of 10 cc Hyaluronic acid gel, in order to prevent postsurgical adhesions.
  Arms: Excision plus hyaluronic acid gel
Procedure: Excision only — Excision of endometriosis foci by laparoscopic standard methods only.
  Arms: Excision only

SUMMARY:
Endometriosis is a common disease of women in the reproductive age and is an important cause for female infertility. Endometriosis is often associated with the development of adhesions which further compromises the fertility of the affected women. The main purpose of this study is to investigate the pregnancy rate one year after excision of endometriosis and application of GnRH-analogues (Gonadotropin-releasing hormone) for 3 month. Half of the patients will receive traditional endometriosis treatment with the excision of the endometriotic lesions only. The other half will additionally receive a gel which can reduce adhesion formation (Hyalobarrier®). Further study objective is the investigation in the development of different types of endometriosis-associated pain over a period of one year. Potential study participants are women with endometriosis-associated pain and with a desire to have children. It will be investigated in the study if the use of Hyalobarrier® will result in a higher pregnancy rate due to reduced adhesion development.

DETAILED DESCRIPTION:
Design: Prospective, monocentric, comparative, randomized, semi-blind.

There will be 30 subjects in each arm, who will be followed 15 months after surgery.

Half of the patients will receive standard laparoscopic excision of the endometriotic lesions only. The other half, after the excision of the endometriosis foci, will receive 10 cc of an antiadhesion agent which contents hyaluronic acid gel (Hyalobarrier®).The subjects will be hospitalized after surgery for at least 2 days.

A Vas-Scala will be given to the subjects to estimate the pain before, after surgery and one year after treatment. The participants will record the values each three months after surgery.

All subjects will be asked by telephone for the VAS-scala values and for pregnancy (Date of Initiation, clinical evolution)

The participation ist voluntary and an Informed consent must be signed before surgery. Subjects are free to withdraw their consent anytime.

ELIGIBILITY:
Inclusion Criteria:

* Women over 18 years with endometriosis-associated pain, like dysmenorrhea, dyspareunia, lower abdominal pain, low-back pain, rectal pain, defecation pain (only one criterion needs to be fulfilled for study inclusion);
* Participants are in good general health except for endometriosis related problems;
* Except for endometriosis, no existence of an obvious diseases which could cause chronic pain or which could cause abdominal pain;
* The participant must have a desire to have children;
* Participants must be able to give their consent and must understand the risks associated with a participation in the study;
* There must be a signed and dated informed consent which was accepted by the local ethic committee

Exclusion Criteria:

* Existent pregnancy including ectopic pregnancy;
* Identification of other causes for the discomfort;
* Chronic diseases, except endometriosis, which require continuous pain therapy;
* Previous application of GnRH analogues 6 month prior to study;
* Concurrent use of systemic corticosteroids, antineoplastic agents and/or radiation;
* Planned additional general surgical procedures during the operation for removal of the endometriotic lesions;
* Absence of endometriosis at laparoscopy;
* Partial resection of the bowel or urinary bladder for removal of endometriosis

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2015-05; Primary Completion 2017-05 (Estimated); Study Completion 2017-05 (Estimated)

PRIMARY OUTCOMES:
Pregnancy rate | One year after completion of endometriosis treatment (excision followed by 3 month of GnRH-analogues)

SECONDARY OUTCOMES:
Endometriosis-associated pain | The day before laparoscopy is performed
  Outcome measure is measured by visual analogue scale
Endometriosis-associated pain | One year after completion of endometriosis treatment
  Outcome measure is measured by visual analogue scale

CONTACTS AND LOCATIONS:
Overall Officials: Rudy L De Wilde, Professor, Principal Investigator — Pius-Hospital Oldenburg, Department of Gynecology, Obstetrics and Gynecological Oncology
Locations (1):
- Pius-Hospital, Department of Gynecology, Obstetrics and Gynecological Oncology, Carl von Ossietzky University, Oldenburg, Lower Saxony, Germany